CLINICAL TRIAL: NCT04712682
Title: Factors Affecting Neck Posture in Academicians With Non-specific Neck Pain
Status: Completed | Type: Observational
Sponsor: Atılım University (Other)
Responsible Party: Principal Investigator, NAİME ULUG, assistant professor, Atılım University
Other Study IDs: 59394181-604.01.01-752
Record Dates: First submitted 2020-10-19; First posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Craniovertebral Angle; Neck Pain; Work-Related Condition
Keywords: craniovertebral angle; Neck Pain; Work-Related Condition
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Assessment of neck posture. — pain, pain threshold, CVA angle, muscle strenght test, joint position sense test

SUMMARY:
There is evidence showing that musculoskeletal problems in the cervical and thoracic region are common among academicians and with it, compared to other musculoskeletal pain the pattern and physical risk factors for neck pain was at the highest percentage.

One of the most common postural disorders in the neck and shoulder girdle occurs when the position of the head is displaced to forward relation to the point of support, which is called forward head posture (FHP).

The aim of the present study is to investigate factors affecting neck posture in academicians with non-specific neck pain.

Investigators investigated whether there is a correlation between craniovertebral angle (CVA) and joint position sense, deep cervical muscle strength and endurance in academicians with chronic non-specific neck pain.

DETAILED DESCRIPTION:
Chronic non-specific neck pain is one of the most important common musculoskeletal problem which has considerable impact on personal and financial costs. Because of physical work factors, neck pain is significantly associated with holding the neck in a prolonged forward posture and performing repetitive movements.

Proper posture is deﬁned as a musculoskeletal balance which involves a minimal amount of stress and strain on the body. Postural assessment is one of the most important parts of the physical examination process. Although correct posture is desired, many people do not exhibit good posture.

Forward head posture(FHP) is the most common cervical postural fault in the sagittal plane that is found with different severity levels in almost all populations.

One of the most common postural disorders in the neck and shoulder girdle occurs when the position of the head is displaced to forward relation to the point of support, which is called forward head posture (FHP). The craniovertebral angle (CVA) is a widely used method for the objective measurement of FHP severity. A smaller CVA indicated a greater FHP and a CVA less than 48-50 is defined as FHP .

It has been reported that approximately 61.3% of adults who work using a computer and have neck pain have an anterior tilt posture of the head. This postural disorder is caused by various factors like sleeping with the head too high, prolonged computer use, weak back muscles, etc. In recent years, the widespread use of computers in offices has caused people to use their personal computers too much in their daily life. These changes can cause a bad posture and accompanying neck pain.

Long-term work in front of a computer requires a static posture of the upper body. To maintain the static posture, the neck, shoulder and upper extremity muscles are overloaded and consequently injured. Uncomfortable posture, especially depending on the viewing angle of the screen and the position of the chair and table, can shorten soft tissues and cause muscle tension, weakness and muscle fatigue. Some researchers reported that the muscle tension and stress that occurs in shortened structures, this condition can cause pain and this can develop a vicious cycle of muscle tension-pain-increased tension-increased pain.

From the point of view of biomechanics, FHP causes changes in the muscle tendon unit length of the cervical extensors and flexors and the atlanto-occipital joint.

The tendency to stay seated for long periods of time is increasing as is the percentage of the population that use a personal computer or smart phone.

This can cause changes in the alignment of the spine, leading to improper posture, such as a rounded shoulder or forward head posture (FHP) . The CVA is a widely used method for the objective measurement of FHP.

The cervical vertebra plays role in proprioceptive sensory input. The proprioceptive perception of the cervical vertebra carry information to correct malalignment and has an important role in postural control. It also reacts sensitively for proper movement of the head by acting in coordination with the sensory feedback from the vestibular system.

FHP can produce problems such as increasing stress on the posterior cervical elements, restriction in range of cervical motion, muscular activity level and impair cervical proprioception.

Academicians may have to be standing position for a long time, use a computer in a static posture, and work in a stressful mood caused by academic progress anxieties.

Accordingly, in a study the academicians reported the upper back and neck regions, as most common musculoskeletal problems.

Researchers found that in academicians compared to other musculoskeletal pain the pattern and physical risk factors for neck pain was at the highest percentage.

To our knowledge, there is no study evaluating factors affecting neck posture in academicians with non-specific neck pain.

The aim of our study is to examine the relationship between neck posture and neck pain and the factors affecting neck posture among academicians.

ELIGIBILITY:
Inclusion Criteria:

* suffering from chronic neck pain greater than 3 months' duration, participated in the study.

Exclusion Criteria:

* diagnosis of cervical radiculopathy or myelopathy and history of cervical and thoracic spine fracture or surgery.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fifty volunteer individual from academic staff diagnosed with nonspecific chronic neck-pain patients agedbetween 22 and 65 years
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2020-06-18 (Actual); Study Completion 2020-07-22 (Actual)

PRIMARY OUTCOMES:
Factors Affecting Neck Posture | 6months
  to investigate if there is a correlation between craniovertebral angle and joint position sense, deep cervical muscle strength and endurance in academicians with chronic non-specific neck pain

CONTACTS AND LOCATIONS:
Locations (1):
- Naime Ulug, Ankara, Select State, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hoy DG, Protani M, De R, Buchbinder R. The epidemiology of neck pain. Best Pract Res Clin Rheumatol. 2010 Dec;24(6):783-92. doi: 10.1016/j.berh.2011.01.019. PMID 21665126
- [Background] Cagnie B, Danneels L, Van Tiggelen D, De Loose V, Cambier D. Individual and work related risk factors for neck pain among office workers: a cross sectional study. Eur Spine J. 2007 May;16(5):679-86. doi: 10.1007/s00586-006-0269-7. Epub 2006 Dec 8. PMID 17160393
- [Background] Haughie LJ, Fiebert IM, Roach KE (1995) Relationship of forward head posture and cervical backward bending to neck pain. J Manual Manip Ther 3(3):91-97
- [Background] Yip CH, Chiu TT, Poon AT. The relationship between head posture and severity and disability of patients with neck pain. Man Ther. 2008 May;13(2):148-54. doi: 10.1016/j.math.2006.11.002. Epub 2007 Mar 23. PMID 17368075
- [Background] Patwardhan AG, Havey RM, Khayatzadeh S, Muriuki MG, Voronov LI, Carandang G, Nguyen NL, Ghanayem AJ, Schuit D, Patel AA, Smith ZA, Sears W. Postural Consequences of Cervical Sagittal Imbalance: A Novel Laboratory Model. Spine (Phila Pa 1976). 2015 Jun 1;40(11):783-92. doi: 10.1097/BRS.0000000000000877. PMID 25768685
- [Background] Nejati P, Lotfian S, Moezy A, Nejati M. The study of correlation between forward head posture and neck pain in Iranian office workers. Int J Occup Med Environ Health. 2015;28(2):295-303. doi: 10.13075/ijomeh.1896.00352. PMID 26182924
- [Background] Khayatzadeh S, Kalmanson OA, Schuit D, Havey RM, Voronov LI, Ghanayem AJ, Patwardhan AG. Cervical Spine Muscle-Tendon Unit Length Differences Between Neutral and Forward Head Postures: Biomechanical Study Using Human Cadaveric Specimens. Phys Ther. 2017 Jul 1;97(7):756-766. doi: 10.1093/ptj/pzx040. PMID 28444241
- [Background] Sauter SL, Schleifer LM, Knutson SJ. Work posture, workstation design, and musculoskeletal discomfort in a VDT data entry task. Hum Factors. 1991 Apr;33(2):151-67. doi: 10.1177/001872089103300203. PMID 1860702
- [Background] Eltayeb S, Staal JB, Hassan A, de Bie RA. Work related risk factors for neck, shoulder and arms complaints: a cohort study among Dutch computer office workers. J Occup Rehabil. 2009 Dec;19(4):315-22. doi: 10.1007/s10926-009-9196-x. PMID 19685174
- [Background] Larsson B, Sogaard K, Rosendal L. Work related neck-shoulder pain: a review on magnitude, risk factors, biochemical characteristics, clinical picture and preventive interventions. Best Pract Res Clin Rheumatol. 2007 Jun;21(3):447-63. doi: 10.1016/j.berh.2007.02.015. PMID 17602993
- [Background] Kang JH, Park RY, Lee SJ, Kim JY, Yoon SR, Jung KI. The effect of the forward head posture on postural balance in long time computer based worker. Ann Rehabil Med. 2012 Feb;36(1):98-104. doi: 10.5535/arm.2012.36.1.98. Epub 2012 Feb 29. PMID 22506241
- [Background] Shaghayegh Fard B, Ahmadi A, Maroufi N, Sarrafzadeh J. Evaluation of forward head posture in sitting and standing positions. Eur Spine J. 2016 Nov;25(11):3577-3582. doi: 10.1007/s00586-015-4254-x. Epub 2015 Oct 17. PMID 26476717
- [Background] Johnson MB, Van Emmerik R EA. Effect of head orientation on postural control during upright stance and forward lean. Motor Control. 2012 Jan;16(1):81-93. doi: 10.1123/mcj.16.1.81. PMID 22402222
- [Background] Ghamkhar L, Kahlaee AH. Is forward head posture relevant to cervical muscles performance and neck pain? A case-control study. Braz J Phys Ther. 2019 Jul-Aug;23(4):346-354. doi: 10.1016/j.bjpt.2018.08.007. Epub 2018 Aug 22. PMID 30145129
- [Background] 15. Basakçı ÇB, Telli AB, Bas ̧gan E, Gökçe B. Analyzing muscu- loskeletal system discomfort, work interference and risk fac- tors of office workers with computer users. Journal of Mar- mara University Institute of Health Sciences. 2013; 3(4): 208- 214.
- [Background] Ozdinc S, Kayabinar E, Ozen T, Turan FN, Yilmaz S. Musculoskeletal problems in academicians and related factors in Turkey. J Back Musculoskelet Rehabil. 2019;32(6):833-839. doi: 10.3233/BMR-181171. PMID 31403936
- [Background] Mohan V, Justine M, Jagannathan M, Bt Aminudin S, Bt Johari SH. Preliminary study of the patterns and physical risk factors of work-related musculoskeletal disorders among academicians in a higher learning institute. J Orthop Sci. 2015 Mar;20(2):410-7. doi: 10.1007/s00776-014-0682-4. Epub 2014 Dec 27. PMID 25542222